CLINICAL TRIAL: NCT02696759
Title: The Gut Microbiome and Gastrointestinal Toxicities as Determinants of the Response to Neoadjuvant Chemotherapies for Advanced Breast Cancer
Brief Title: Gut Microbiome & Gastrointestinal Toxicities as Determinants of Response to Neoadjuvant Chemo for Advanced Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution in 2019. Study was placed on hold at that time and will not be resuming. No data analysis was performed.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 204897
Record Dates: First submitted 2016-02-04; First posted 2016-03-02 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood & Fecal Collection (Other): Subjects receiving neoadjuvant chemotherapy for advanced breast cancer will be asked to complete questionnaires, provide two blood samples, and provide 2 fecal samples while receiving standard of care neoadjuvant chemotherapy
  Interventions: Other: Blood & Fecal Collection

INTERVENTIONS:
Other: Blood & Fecal Collection — Prior to first dose of chemotherapy: (a) Blood sample for research; (b) Fecal sample for research using a kit provided by the research staff for home collection of the fecal sample. The kit may be brought back to the clinic or mailed in a discreet package; (c) Questionnaire on health related quality of life. During chemotherapy: Questionnaires on health related quality of life and regarding any treatment side effects. Questionnaires will be completed every 2 weeks during standard office visits. After chemotherapy, prior to surgery: (a) Blood sample for research; (b) Fecal sample for research using a kit provided by the research staff for home collection of the fecal sample. The kit may be brought back to the clinic or mailed in a discreet package.

SUMMARY:
The purpose of this research is to test whether bacteria that normally live in the intestines play a role in fighting cancer. It is believed that the development and behavior of these immune cells may be influenced by bacteria and other microorganisms living in the gut. In turn, the activities of these immune cells could work with anti-cancer therapies to make them more, or less, effective.

DETAILED DESCRIPTION:
Many chemotherapeutic agents compromise the integrity of the mucosal barrier in the gut, allowing translocation of gram-positive bacteria in secondary lymphoid organs. While this has, until recently, been considered an undesirable side-effect, it may also represent one mechanism by which chemotherapy stimulates an effective anti-cancer immune response. The purpose of this research is to test whether bacteria that normally live in the intestines play a role in fighting cancer. It is believed that the development and behavior of these immune cells may be influenced by bacteria and other microorganisms living in the gut. In turn, the activities of these immune cells could work with anti-cancer therapies to make them more, or less, effective. The hypothesis is that gut microbial composition can influence immune response to the tumor, resulting in inter-individual differences in the response to anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with invasive breast cancer and prescribed a regimen that includes neo-adjuvant therapy prior to breast surgery.
* Able to provide informed consent.

Exclusion Criteria:

* History of previous malignancy, other than non-melanoma skin cancers
* Inability to tolerate phlebotomy
* Immunosuppressive therapy for any other condition
* Fever or active uncontrolled infection in the last 4 weeks
* Inflammatory bowel disease
* Surgery of the stomach, small or large intestines, appendectomy, gastric bypass or gastric banding in the past 6 months.
* Active autoimmune disease, including, but not limited to, Systemic lupus erythematosus (SLE), Multiple sclerosis (MS), ankylosing spondylitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Makhoul, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be shared internally at the University of Arkansas for Medical Sciences (UAMS) or in an National Institutes of Health (NIH)-designated data repository in a manner consistent with all applicable federal and state laws. Subjects who agree to participate in this study, will be given the option to have their data shared; however, opting not to participate in data sharing will have no impact on their study participation.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blood & Fecal Collection
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blood & Fecal Collection
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 53 [32 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Complete Fecal Collection
Description: At least one fecal kit collected
Time Frame: Through study completion, an average of 18 months
Population: Study was halted prematurely. Data analysis not complete.
Measure: Number; unit: participants
Arm/Group | Blood & Fecal Collection
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Blood & Fecal Collection
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The secondary objectives were removed because it was decided (due to a number of parameters including the departure of the PI and failure to meet the enrollment goal) that the samples would not be analyzed. Thus, the secondary objectives in the previous submissions are no longer relevant, and there are no results to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT02696759/Prot_SAP_000.pdf